CLINICAL TRIAL: NCT00400699
Title: UPMC McKeesport/ROCOG Radiation Oncology Minorities Outreach Program
Brief Title: Radiation Therapy Outreach Program for Minority or Low-Income Patients With Newly Diagnosed Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dwight Heron, MD, FACRO, FACR, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PCI-0408108; CDR0000513067 (Registry Identifier: PDQ (Physician Data Query)); NCT00304343 (obsolete NCT alias)
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Psychosocial Effects of Cancer and Its Treatment; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: psychosocial effects of cancer and its treatment; unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Counseling; Psychiatric Rehabilitation

ARMS (1):
- REview (Other)
  Interventions: Other: counseling intervention; Other: study of socioeconomic and demographic variables; Procedure: psychosocial assessment and care

INTERVENTIONS:
Other: counseling intervention
Other: study of socioeconomic and demographic variables
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: An outreach program may help minority or low-income cancer patients overcome problems that keep them from receiving quality care.

PURPOSE: This clinical trial is studying how well a radiation therapy outreach program works in minority or low-income patients with newly diagnosed cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop, over five years, and implement a shared infrastructure that will permit participating community cancer centers to participate in radiation oncology clinical research and dramatically increase their rate of trial accrual above historical patterns.
* Increase access to radiation oncology services and clinical trials for underserved minority and/or low-income patients in the target areas, through community and professional education and outreach activities.
* Assess and ensure the quality of radiation oncology services at participating facilities through the use of a new integrated radiation oncology outcomes database and a quality assurance program, benchmarking daily practice patterns to clinical practice protocol.
* Compare treatment approaches and outcomes for cervical, colorectal, lung, prostate, breast, and head and neck cancers across racial and socioeconomic status groups.
* Conduct community intervention pilot programs that advance the understanding of factors that lead to health disparities.
* Develop and implement clinical treatment studies that attempt to reduce or eliminate health disparities through novel treatment approaches.
* Develop and refine a model program that can be sustained by the community treatment facilities long after study completion, and that the National Cancer Institute or other similarly motivated funders can replicate within other regions.

OUTLINE: This is a multicenter study.

Patients are enrolled in the Patient Navigator program, an initiative to promote equal access and quality of cancer care. Patients undergo an interview with the Patient Navigator, who is an oncology health professional, over approximately 1 hour to identify specific needs, in terms of receiving cancer care. The interview serves as a basis for developing a plan to assist patients through treatment and follow up. The Patient Navigator meets the patient, in person or over the phone, at various times during treatment to help the patient overcome barriers to completion of cancer therapy. The Patient Navigator then provides yearly follow up to facilitate continued medical follow up. Patients complete surveys before and after program participation.

Patients are followed periodically to determine their current status in cancer therapy.

TELESYNERGY®, a portable live-time interactive telemedicine system, is utilized in developing the necessary infrastructure and professional education in the community. It is used for sharing information and approaches for case presentation, treatment planning conferences, and other specialized presentations by invited speakers and expert panels. Activities using the TELESYNERGY® system are videotaped to create a library of topic-centered presentations that can be shared with the larger community. Components and summaries are placed on an Internet site to encourage communication with the larger oncology community.

PROJECTED ACCRUAL: A total of 3,150 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed cancer
* Receiving radiation therapy and/or chemotherapy
* Minority and/or economically disadvantaged population

PATIENT CHARACTERISTICS:

* Within any of the following service areas of 5 different hospitals in western Pennsylvania:

  * New Castle
  * Pittsburgh Metro
  * Somerset
  * Mckeesport
  * Johnstown
* Any race, ethnicity, gender, or HIV status allowed

  * HIV serostatus is not evaluated specifically for study participation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3150 (Actual)
Dates: Start 2004-10; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Clinical stage at time of presentation (indicator of early access to system) | Observation
Date and nature of post-diagnosis surgery or biopsy | Observation
Proportion of patients compliant with treatment plan | Observation
Total radiation dosage per patient (curative and palliative endpoints) | Observation
Supportive services provided to patients | Observation
Rate of treatment completion | Observation
Accrual for clinical research protocols | Observation
Retention in clinical research protocols | Observation
Barriers to treatment (perceived and real) | Observation

CONTACTS AND LOCATIONS:
Overall Officials: Dwight E. Heron, MD, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Cancer Center - New Castle, New Castle, Pennsylvania
  - Mercy Cancer Institute at Mercy Hospital, Pittsburgh, Pennsylvania
  - Somerset Oncology Center, Somerset, Pennsylvania